CLINICAL TRIAL: NCT03770221
Title: Coordinating Access to Care for People Experiencing Homelessness: The Role and Impact of Financial Incentives
Brief Title: Coordinating Access to Care for People Experiencing Homelessness (CATCH-FI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Collaborators: Ontario Ministry of Health and Long Term Care (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: REB#: 18-196
Record Dates: First submitted 2018-11-05; First posted 2018-12-10 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Mental Health Disorder
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Financial Incentive (Experimental): Participants will receive usual brief, intensive case management to connect them to health and social services and supports in the community.
  Additionally, participants in this arm will receive $20 for every week they maintain contact with CATCH service providers, as required by their care plan. Contact can be by phone, text, email, or in person with CATCH service providers over 6 months of follow up, or until they are successfully transitioned to longer-term supports (for up to $80/month per participant).
  Interventions: Behavioral: CATCH; Other: Financial Incentive
- Usual Care (Active Comparator): Participants will receive usual brief, intensive case management to connect them to health and social services and supports in the community.
  Interventions: Behavioral: CATCH

INTERVENTIONS:
Behavioral: CATCH — Brief, intensive case management service.
  Other Names: Coordinated Access to Care for the Homeless
Other: Financial Incentive — Financial incentive for maintaining contact with CATCH service providers.
  Arms: Financial Incentive

SUMMARY:
Coordinating Access to Care for the Homeless (CATCH) initiative is a multidisciplinary brief intervention for homeless adults with mental health needs discharged from hospital in Toronto, Canada. The study aims to evaluate the effect of financial incentives in facilitating treatment engagement of homeless people with mental illness, as well as in improving health, health service use and housing outcomes, compared to usual CATCH care, over 6 months, a critical time of transition from hospital to community care.

ELIGIBILITY:
Inclusion Criteria:

* able to give informed consent
* a new client of the CATCH team, recently admitted or readmitted
* at least one contact with the CATCH team

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2018-11-19 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Number of contacts with CATCH service providers | 6 months
  The number of contacts (per month) with CATCH service providers (established by review of program records) until the transition to long-term care providers is accomplished.

SECONDARY OUTCOMES:
Number of hospitalizations | 1 year prior to enrolment, 1 year post-enrolment
  We will establish the number of hospitalizations, during the year prior to program enrolment and the 1 year follow-up period. Data linkage will be conducted at the Institute for Clinical Evaluative Sciences (ICES), where population-based health information is available at the patient level for all Ontarians using formal health services. Health service use will be examined by the National Ambulatory Reporting System (NACRS), the Discharge Abstract Database (DAD), the Ontario Mental Health Reporting System (OMHRS) and the Ontario Health Insurance Plan (OHIP) for ED visits, outpatient clinics, and inpatient hospitalizations. The project will attain health service data for all consenting participants from 12 months prior to study enrolment to 12 months following study enrolment.
Days in hospital | 1 year prior to enrolment, 1 year post-enrolment
  We will establish the number of days is hospital during the year prior to program enrolment and the 1 year follow-up period. Data linkage will be conducted at the Institute for Clinical Evaluative Sciences (ICES), where population-based health information is available at the patient level for all Ontarians using formal health services. Health service use will be examined by the National Ambulatory Reporting System (NACRS), the Discharge Abstract Database (DAD), the Ontario Mental Health Reporting System (OMHRS) and the Ontario Health Insurance Plan (OHIP) for ED visits, outpatient clinics, and inpatient hospitalizations. The project will attain health service data for all consenting participants from 12 months prior to study enrolment to 12 months following study enrolment.
Number of emergency department visits | 1 year prior to enrolment, 1 year post-enrolment
  We will establish the number of emergency department visits during the year prior to program enrolment and the 1 year follow-up period. Data linkage will be conducted at the Institute for Clinical Evaluative Sciences (ICES), where population-based health information is available at the patient level for all Ontarians using formal health services. Health service use will be examined by the National Ambulatory Reporting System (NACRS), the Discharge Abstract Database (DAD), the Ontario Mental Health Reporting System (OMHRS) and the Ontario Health Insurance Plan (OHIP) for ED visits, outpatient clinics, and inpatient hospitalizations. The project will attain health service data for all consenting participants from 12 months prior to study enrolment to 12 months following study enrolment.
Mental health symptom severity | Baseline, 6 months
  The Colorado Symptom Index (CSI) was designed specifically for homeless individuals with mental health problems. It is a 14-item instrument which assesses the presence and frequency of symptoms of mental illness experienced within the past month. Responses are provided using a 5-point Likert scale with answer choices ranging from 0 (not at all) to 4 (at least every day). A higher score indicates a higher level of symptoms. The CSI is a widely used tool in research as a self-report measure of psychiatric symptomatology. The CSI has been reported to have excellent internal consistency (.92) and test-retest reliability (.71). Evidence of the CSI's validity is strong as CSI scores have been proven to distinguish between individuals with and without mental health service needs and were significantly correlated with functioning.
Health status | Baseline, 6 months
  The Short Form 36 (SF-36) 36-item self-report measure of generic health status is designed to produce Physical Component Summary (PCS) and Mental Component Summary (MCS) scores. There are scaled questions concerning physical functioning, role limitations, bodily pain, general health perceptions, vitality, social functioning, and general mental health (psychological distress and psychological well-being). Each scale is directly transformed into a 0-100 scale, with lower scores indicating poorer health status. SF-36 has excellent psychometric properties and has been used successfully in a variety of settings and diagnostic groups, including the homeless population.
Working Alliance | 6 months
  Participants will be asked to complete the 12-item Working Alliance Inventory - Short Revised (WAI-SR) questionnaire, to assess how they think and feel about the therapeutic relationship with their case manager. Responses are provided using a 5 point Likert scale ranging from 1 (Seldom) to 5 (Always).The WAI-SR includes three subscales relating to task, goal, and bond, and yields a summary score that ranges from 12 to 60, with higher scores indicating a stronger therapeutic relationship.
Substance use | Baseline, 6 months
  The Global Appraisal of Individual Needs Short Screener (GAIN-SS), extensively used in this population, consists of questions on four subscales: internal distress, external distress, substance distress, and crime/violence . Response options are: in the 'past month' =4, '2-3 Months'=3, '4-12 Months' =2, or '1+ years.'=1, or 'Never'=0. Using these questions, the GAIN past month score is calculated by counting the number of times the participant identified that they had these problems in the last month, with a higher score indicating greater severity of substance use problems. Scores have 3 levels of severity including: Low (0), Moderate (1 to 2) and High (3+). In addition, we will elicit information on the number of days in the 30 days that participants have problems with alcohol or drugs, and the amount of money spent on alcohol or drugs in the past 30 days.
Housing stability | Baseline, 6 months
  This modified version of the Dartmouth Residential Time-Line Follow-Back (RTLFB) is designed to collect detailed information about a participant's type of housing and number of days stably housed. The RTFLB uses a calendar and prompts to collect housing for specific time periods. In this study, this information will inform questions about housing stability and circumstances and is being collected at baseline and 6 months. The outcome of interest is the number of days stably housed in the past 6 months.
Disease-Specific Quality of Life: Lehman Quality of Life scale | Baseline, 6 months
  The original Lehman Quality of Life scale was designed to assess the quality of life of people with severe mental illness. It is a structured self-report interview, conducted by a trained non-clinical interviewer, and elicits participants' ratings of their quality of life. There are 7 subjective scales (living situation, everyday activities, family, social relationships, finances, safety, and satisfaction with life in general) and 4 objective scales (everyday activities, enough money, family contacts, and contacts with friends), scored on a Likert scale ranging from Terrible=1 to Delighted=7. A higher score indicates a higher quality of life. This shorter 20-item version (QoLi-20) was developed and validated by Uttaro and Lehman and used extensively in the homeless population.
Health-related quality of life: EQ-5D-5L | Baseline, 6 months
  The EuroQol-5Dimensions-5Levels (EQ-5D-5L) is a generic measure of health-related quality of life. The EQ-5D-5L includes five items concerning mobility, self-care, usual activities, pain/discomfort, and anxiety/depression that are weighted(on a scale ranging from Level 1, indicating no problem, to Level 5, indicating extreme problems) to produce a single utility score between 0 and 1. The Visual Analogue Scale (VAS) of the EQ-5D will also be included, which will allow participants to rate their overall health, mental health and physical health from 0 to 100, where a higher score indicates better overall health.
Income support | Baseline, 6 months
  Participants will be asked to provide their income for the previous month from a number of sources, including: all jobs, Ontario Works, Ontario Disability Support Program, Employment Insurance, child benefits, child support, all other sources of income (pensions, investments, Trillium benefits, HST rebates, etc.).

CONTACTS AND LOCATIONS:
Overall Officials: Vicky Stergiopoulos, MD, MHSc, Principal Investigator — Unity Health Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Reid N, Nisenbaum R, Hwang SW, Durbin A, Kozloff N, Wang R, Stergiopoulos V. The Impact of Financial Incentives on Service Engagement Among Adults Experiencing Homelessness and Mental Illness: A Pragmatic Trial Protocol. Front Psychiatry. 2021 Aug 3;12:722485. doi: 10.3389/fpsyt.2021.722485. eCollection 2021. PMID 34413804